CLINICAL TRIAL: NCT05419258
Title: Feasibility and Evaluation Study of the UPLUG Hemodialysis Connection Device
Acronym: UPLUG-SAFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 21-0265
Record Dates: First submitted 2022-04-29; First posted 2022-06-15 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2023-07

CONDITIONS: Hemodialysis; Renal Insufficiency, Chronic
Keywords: medical device; connection medical device
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: feasibility study on medical device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- use of the device during hemodialysis sessions (Experimental): use of the device during one month during hemodialysis sessions
  Interventions: Device: UPLUG Hemodialysis Connection Device

INTERVENTIONS:
Device: UPLUG Hemodialysis Connection Device — use of the device UPLUG during 1 month

SUMMARY:
The new Uplug° technology, interface between the end of the hemodialysis catheter and the dialysis circuit, makes it possible to limit direct access to the hemodialysis catheter during connections and disconnections.

Aim:

The investigators propose a feasibility study, in order to study the new Uplug° technology in real conditions of use.

Material and methods:

This study aim to include 15 hemodialysis patients in a center on a tunneled permanent central venous hemodialysis catheter. The Uplug° technology will be placed at the end of each patient's hemodialysis catheter for a period of one month.

Hypothesis tested:

The main endpoint is the proportion of hemodialysis sessions performed successfully with this technology, respecting the usual dialysis prescription.

DETAILED DESCRIPTION:
The incidence and prevalence of chronic insufficiency have been growing for several years. Increasingly older patients are treated with chronic hemodialysis. The vascular access of choice remains the arteriovenous fistula and the proportion of hemodialysis patients on the permanent central venous hemodialysis catheter varies from 20 to 35% in dialysis centres. The new Uplug° technology, interface between the end of the hemodialysis catheter and the dialysis circuit, makes it possible to limit direct access to the hemodialysis catheter during connections and disconnections.

Aim:

The investigators propose a feasibility study, in order to study the new Uplug° technology in real conditions of use.

Material and methods:

This study aim to include 15 hemodialysis patients in a center on a tunneled permanent central venous hemodialysis catheter. The inclusion period is three months. The follow-up time for each participant is 6 weeks. Patients with a tunneled permanent central venous hemodialysis catheter and performing dialysis sessions with a flow rate ≥ 300 ml/min may be included. The Uplug° technology will be placed at the end of each patient's hemodialysis catheter for a period of one month.

Hypothesis tested:

The main endpoint is the proportion of hemodialysis sessions performed successfully with this technology, respecting the usual dialysis prescription.

The secondary objectives are the infectious risk, the defects of the experimental device and the hemodialysis catheter or their implementation, the satisfaction of the nursing staff and the patient, the reduction in the number of manipulations and the effective time of these manipulations.

ELIGIBILITY:
Inclusion Criteria:

* with end-stage chronic renal failure treated by hemodialysis (2 or 3 sessions per week)
* Wearer of a right or left jugular permanent tunneled central venous hemodialysis catheter whose end has been in the superior vena cava or the right atrium for at least 1 month
* Hemodialysis catheter lock used = heparin or 4% citrate
* Expected life expectancy > 6 months
* Dialysis session preceding inclusion with an average blood flow of at least 300ml/min

Exclusion Criteria:

* Patient with a mechanical heart valve
* Patient with an arteriovenous fistula (AVF) that can be used within one month
* Kidney transplant by living donor planned in the following month
* Pregnant or breastfeeding woman
* History of infection on the hemodialysis catheter in place dating from less than 6 months
* Psychiatric or demented patient unable to obtain informed consent
* Patient already included in another protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
success in performing dialysis | one month
  Study the feasibility of performing dialysis with the UPlug Technology in patients with a permanent tunneled central venous hemodialysis catheter with the objective of a success rate ≥ 80%.

SECONDARY OUTCOMES:
Number of participants with Adverse Events [Safety and Tolerability] of the experimental device UPLUG | one month
  adverse events reported from consent to end of study
experimental device integrity | one month
  device deficiencies reported from consent to end of study
nurses' satisfaction | one month
  satisfaction evaluated by questionnaire before and after the inclusions
patient satisfaction | one month
  satisfaction evaluated by questionnaire before and after the use of experimental device
clinical performance of device | one month
  performance measured by rate of successful sessions

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen Normandie, Caen, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR